CLINICAL TRIAL: NCT06900816
Title: A Single-centre, Single-dose, Open Label, Non-randomized, Parallel Group, Clinical Pharmacology Study of CHF 6001 in Asthmatic Adolescent Patients and in Asthmatic Adult Patients as Control Group
Brief Title: A Comparison Study Between Adolescents With Asthma and Adults With Asthma on How They Absorb, Metabolise and Eliminate CHF 6001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLI-06001AC1-01; 2024-516483-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-03-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: CHF6001; pharmacokinetics; adolescents; patients
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- adolescent patients (Experimental): CHF 6001 dry powder inhaler (DPI) device, followed by a safety follow-up visit be done 12 to 14 days after the subject's study treatment administration. There is no comparator and all patients will receive the same study treatment.
  Interventions: Drug: CHF 6001
- Adult patients (Experimental): CHF 6001 dry powder inhaler (DPI) device, followed by a safety follow-up visit be done 12 to 14 days after the subject's study treatment administration. There is no comparator and all patients will receive the same study treatment.
  Interventions: Drug: CHF 6001

INTERVENTIONS:
Drug: CHF 6001 — CHF 6001 DPI single dose
  Arms: adolescent patients
Drug: CHF 6001 — CHF 6001 DPI single dose
  Arms: Adult patients

SUMMARY:
The purpose of this study is to evaluate the amount of the study drug, CHF6001, in the blood of adolescent patients with asthma in comparison to adult patients with asthma after a single oral dose of the study drug, CHF 6001.

DETAILED DESCRIPTION:
The study plan foresees a total of four visits at clinic. At Visit 1, after the signature of the informed consent form, the inclusion/exclusion criteria will be checked and the lung function parameters will be evaluated. If the subjects meet the inclusion/exclusion criteria, they will be trained to assess their ability to use an inhaler device and to teach the inhaling technique. At the following visit, the patients will inhale through the device and amount of the study drug and of its metabolites in the blood will be measured at different times after inhalation. At a subsequent ambulatory visit, the final measurements will be performed. A follow-up Visit will be done to check patients safety and wellbeing, 12 to 14 days after the study treatment intake. A total of 25 asthmatic adults (≥18 years), and 25 asthmatic adolescents ( ≥12 and <18 years) with a stable asthma therapy according to international guidelines Global Initiative for Asthma (GINA) (update 2024), will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: subject's and/or parents or legal representative (for adolescents) written informed consent obtained prior to any study-related procedures.
2. Sex and age: a. Adolescent: male or female subjects aged ≥12 and <18 years; b. Adult: male or female subjects aged ≥18 and ≤75 years.
3. Body weight for adolescents within the range of ≥34.7 kg for 12 years old and ≥40.4 kg for 13 to 17 years old.
4. Body mass index for adults within the range of ≥18.0 to ≤30.0 kg/m2.
5. Diagnosis of asthma: a documented history of physician diagnosed asthma according to international guidelines (GINA) update 2024 for ≥1 year, with diagnosis before the age of 50 years for adults.
6. Stable asthma therapy: a stable treatment with medium dose of inhaled corticosteroids (ICS) (medium-dose ICS defined as beclometasone dipropionate [BDP] non-extrafine >500 to 1000 μg or estimated clinical comparable dose as per GINA guidelines update 2024) alone or in fixed combination with a Long-acting β2-agonist (LABA) with or without long-acting muscarinic antagonist (for subjects ≥18 years old only) for ≥3 months before screening.
7. Lung function: adolescent and adult subjects with a Forced Expiratory Volume in 1 Second (FEV1) >70% of predicted values (% predicted) after withholding short-acting β2-agonist (SABA) treatment for a minimum of 6 hours before screening or 24 hours in case of ICS and LABA (alone or in fixed combination).
8. A cooperative attitude and ability: a. To correctly use the inhalers; b. To perform all study-related procedures including technically acceptable spirometry according to the 2019 American Thoracic Society (ATS)/ European Respiratory Society (ERS) guidelines.
9. Female subjects fulfilling one of the following criteria: a. Women of non-childbearing potential (WONCBP) defined as physiologically incapable of becoming pregnant (i.e., postmenopausal or permanently sterile, as per definitions given in Section 1.1 of the Clinical Trials Coordination Group (CTCG) guidance). Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per Investigator's request, postmenopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges). b. Women of childbearing potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up (FU) visit or; ii. WOCBP with non-fertile male partners (contraception is not required in this case). For the definition of WOCBP, fertile men and the list of highly effective birth control methods, refer to or Section 1.1 and 4.1 of the CTCG guidance.

Exclusion Criteria:

1. Blood donation (≥450 mL) or blood loss, less than 2 months before screening or before enrolment on Day 1, applicable for adults only.
2. History of "at risk" asthma: history of near fatal asthma or of a past hospitalisation for asthma in intensive care unit which, in the judgement of the Investigator, may place the subject at undue risk.
3. Recent exacerbation or respiratory tract infection: hospitalisation, emergency room admission or use of systemic corticosteroids for an asthma exacerbation or respiratory tract infection in the 4 weeks before the screening visit. Note: Subjects experiencing an exacerbation or respiratory tract infection during the screening visit may be rescreened once, ≥6 weeks after recovery. If there is no recovery, such event constitutes an exclusion criterion and leads to screening failure.
4. Subjects using systemic corticosteroid medication 4 weeks or slow release corticosteroids 12 weeks before enrolment.
5. Patients being treated with anti-inflammatory asthma monoclonal antibodies or biological drugs which can affect asthma inflammation within 6 months before or five half-lives (whichever is greater) before the screening visit.
6. Respiratory disorders other than asthma: subjects with known respiratory disorders other than asthma. This can include, but is not limited to, Chronic Obstructive Pulmonary Disease (COPD), α1-antitrypsin deficiency, active tuberculosis, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease and others.
7. Smoking status: current smoker, ex-smoker with a smoking history of ≥10 pack-years (pack-years = the number of cigarette packs per day times the number of years) or current use of inhaled or oral cannabis products. Ex-smokers must have stopped smoking for ≥1 year (≥6 months for e-cigarettes).
8. Alcohol/drug abuse: subjects with a known or suspected history of alcohol and/or drug abuse within 12 months before screening.
9. Cancer or history of cancer: subjects with active cancer or a history of cancer with <5 years disease free survival time (whether there is evidence of local recurrence or metastases). Localised carcinoma (e.g., basal cell carcinoma, in situ carcinoma of the cervix adequately treated) is acceptable.
10. Cardiovascular disease: subjects who have clinically significant (CS) cardiovascular condition according to Investigator's judgement, such as heart failure (New York Heart Association class >3), acute ischemic heart disease in the last year prior to screening, history of sustained cardiac arrhythmias or sustained and non-sustained cardiac arrhythmias diagnosed in the last 6 months prior to screening (sustained means lasting >30 seconds or ending only with external action, or leads to haemodynamic collapse; nonsustained means >3 beats <30 seconds, and/or ending spontaneously and/or asymptomatic), high degree impulse conduction blocks (>2nd degree atrioventricular block type 2). Similarly, subjects affected by persistent, long-standing or paroxysmal atrial fibrillation will not be considered for enrolment. Note: Subjects with permanent atrial fibrillation (for ≥6 months before the screening visit) with a resting ventricular rate <100/min, controlled with a rate control strategy (i.e., selective β-blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) can be considered for enrolment.
11. Electrocardiogram (ECG) criteria: an abnormal and CS 12-lead ECG that in the Investigator's opinion would affect efficacy or safety evaluation or place the subjects at risk. Male subjects whose 12-lead ECG shows Fridericia's Corrected QT Interval (QTcF )>450 ms or female subjects with a QTcF >460 ms (adolescent females) or >470 ms (adult females) at screening or at enrolment (criterion not applicable for subjects with pacemaker or permanent atrial fibrillation).
12. Other severe acute or chronic medical or malignancy or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
13. Liver diseases: subjects with severe hepatitis, chronic active hepatitis or evidence of uncontrolled chronic liver disease according to the Investigator's opinion.
14. Drugs with hepatoxicity potential: subjects receiving treatment with any drug known to have a well-defined potential for hepatotoxicity (i.e., isoniazide, nimesulide, ketoconazole) and strong inhibitors of cytochrome P450 (CYP) 3A4/5 (i.e., itraconazole) within the previous 3 months before the screening visit.
15. Subjects having received a vaccination within 2 weeks before the screening visit.
16. Subjects with major surgery in the 3 months before the screening visit or planned surgery during the study.
17. Subjects with a history of hypersensitivity and/or idiosyncrasy to any of the test compounds or excipients employed in this study.
18. Subjects treated with monoamine oxidase inhibitors or tricyclic antidepressants.
19. Subjects treated with non-potassium sparing diuretics (unless administered as a fixed dose combination with a potassium conserving drug or changed to potassium sparing agent before the screening), non-selective beta blocking drugs, quinidine, quinidine-like anti-arrhythmics or any medication with a Corrected QT Interval (QTc) prolongation potential or a history of QTc prolongation.
20. Subjects who are receiving any therapy that could interfere with the study treatments according to Investigator's opinion.
21. Subjects who have received an investigational drug within 30 days or five half-lives (whichever is greater) prior to the screening visit, or have been previously randomised in this study or are currently participating in another study.
22. Documented coronavirus disease 2019 diagnosis within the last 2 weeks, or associated complications or symptoms, which have not resolved within 14 days before screening.
23. For females only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive serum human chorionic gonadotropin laboratory test at screening visit and urine test at Day 1.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — biological females and biological males
Enrollment: 50 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CHF 6001 after oral inhalation of CHF 6001 Dry Powder Inhaler (DPI) | Samples will be collected at the following time points: pre dose and post-dose at 30 minutes and 1, 2, 4, 8, 10, 24, 48, 72 and 96 hours
  Measurements are performed to define the Pharmacokinetic (PK) profile after oral inhalation of CHF 6001 DPI in adolescent subjects with asthma in comparison to adult subjects with asthma.
Area under the curve from 0 to the last quantifiable concentration (AUC 0-t) of CHF 6001 after oral inhalation of CHF 6001 DPI | Samples will be collected at the following time points: pre dose and post-dose at 30 minutes and 1, 2, 4, 8, 10, 24, 48, 72 and 96 hours
  Measurements are performed to define the PK profile after oral inhalation of CHF 6001 DPI in adolescent subjects with asthma in comparison to adult subjects with asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Iva Popova, MD, Principal Investigator — MC Comac Medical Ltd.
Locations (1):
- Medical Centre Comac Medical Ltd., Sofia, Krasno Selo District, Bulgaria

IPD SHARING:
Plan to Share IPD: No